CLINICAL TRIAL: NCT06741995
Title: DCM Anti-Heart Antibody Diagnostic Kit Study--assessment of the Prognostic Impact of Anti-beta1AR Antibody and Anti-L-CaC Antibody in Patients With Dilated Cardiomyopathy
Brief Title: Evaluating the Prognostic Impact of Anti-β1AR Antibodies and Anti-L-CaC Antibodies in Patients With Dilated Cardiomyopathy
Status: Recruiting | Type: Observational
Sponsor: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Responsible Party: Sponsor
Other Study IDs: Jing yuan-DCM cohort study
Record Dates: First submitted 2024-12-15; First posted 2024-12-19 (Actual); Last update posted 2025-04-11 (Actual); Status verified 2024-12

CONDITIONS: Dilated Cardiomyopathy (DCM)
MeSH Terms: conditions — Cardiomyopathy, Dilated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples remaining after completion of routine clinical blood tests will be destroyed in accordance with the regulations of the hospitals in which the centers are located. The study doctor will take an additional 5ml of blood sample for AHA testing in addition to the routine clinical blood tests. Prior consent will be obtained from the patients before the blood samples are taken; after the completion of the study, the remaining blood samples from the additional 5 ml of blood samples will be approved by the Ethics Committee and used for future research on the mechanism of the development of DCM according to ethical requirements
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Background of the study The etiology of dilated cardiomyopathy (DCM) is complex and involves a variety of genetic, environmental, and immunologic factors. Autoimmune reactions (especially anti-cardiac autoantibodies) play an important role in the development of DCM. In recent years, several clinical studies have suggested that anti-β1AR and anti-L-CaC antibodies are associated with cardiovascular death, ventricular tachycardia, and sudden death in patients with DCM, which is of great value in the prognostic evaluation of DCM. However, most of these studies are single-center studies with small sample sizes and non-uniform testing methods. In this study, we will use a multicenter, prospective cohort study to follow up DCM patients in China for a period of 3 years, to further accurately assess the clinical predictive value of anti-β1AR antibody and anti-L-CaC antibody on the prognosis of DCM patients, and to provide epidemiological information as well as targeted therapeutic targets for DCM.

Aims of the study A multicenter, prospective cohort study of anti-β1AR and anti-L-CaC antibodies for prognostic assessment of DCM patients, enrolling 1,000 DCM patients, to further accurately assess the prognostic value of the anti-AHA assay for DCM patients, and to provide targets for targeted treatment of DCM.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75, any gender
2. Diagnosed with dilated cardiomyopathy
3. Subjects or their legal guardians are fully informed of the nature and risks of the study, participate voluntarily, and sign an informed consent form.

Exclusion Criteria:

1. Serious uncontrolled infection at enrolment ("uncontrolled" is defined as signs and symptoms of infection that persist without improvement despite antimicrobial or other treatment)
2. Uncontrolled active bleeding at enrollment
3. Pregnancy or breastfeeding
4. Combination of serious diseases affecting survival, such as tumors, with a life expectancy of less than one year
5. Previous heart transplant or implantation of a cardiac assist device
6. Patients with poor compliance who are unable to complete the full course of the study
7. Other conditions (e.g., overstimulation, sensitivity, cognitive impairment, mental illness, or substance abuse/addiction) that, in the judgment of the investigator, may increase the risk to the subject or interfere with the clinical study and judgment of the results.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Dilated cardiomyopathy (DCM) is a heterogeneous cardiomyopathy characterized by ventricular enlargement and reduced myocardial contractile function, with the exception of hypertension, heart valve disease, congenital heart disease, or ischemic heart disease at the onset. The clinical manifestations of dilated cardiomyopathy include progressive cardiac enlargement, reduced ventricular systolic function, heart failure, ventricular or supraventricular arrhythmias, conduction system abnormalities, thromboembolism, and sudden death.The etiology of DCM is complex and involves a variety of factors, including genetics, environment, and immunity.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2024-12-17 (Actual); Primary Completion 2027-12-17 (Estimated); Study Completion 2027-12-17 (Estimated)

PRIMARY OUTCOMES:
Composite Endpoint of All-Cause Death, Heart Transplantation, and Rehospitalization for Heart Failure | End of months 1, 6, 12, 18, 24 and 36

SECONDARY OUTCOMES:
All-cause death, heart transplant, heart failure rehospitalization, or sudden death | End of months 1, 6, 12, 18, 24 and 36

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Cardiology, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, 430022, China, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No